CLINICAL TRIAL: NCT07150169
Title: Individualized Magnetic Stimulation for Post-stroke Cognitive Recovery: Optimization, Validation & Efficacy
Acronym: IMPROVE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jord Vink (Other)
Responsible Party: Sponsor-Investigator, Jord Vink, Principal investigator, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: NL-009409
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: stroke; transcranial magnetic stimulation; cognitive impairment; TMS; TMS disruption; fMRI
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: We will perform a prospective mechanistic sham-controlled crossover intervention study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TMS disruption (Experimental): Active TMS disruption delivered at 110% RMT
  Interventions: Device: Active TMS disruption
- Sham TMS disruption (Sham Comparator): Active TMS disruption delivered at 20% RMT
  Interventions: Device: Sham TMS disruption

INTERVENTIONS:
Device: Active TMS disruption — Active TMS disruption delivered to the personalized target
  Arms: Active TMS disruption
Device: Sham TMS disruption — Sham TMS disruption delivered to the personalized target
  Arms: Sham TMS disruption

SUMMARY:
Rationale: 75% of all stroke survivors suffer from cognitive deficits in the acute phase, with serious implications for their long-term quality of life and societal participation. A promising novel therapy is repetitive transcranial magnetic stimulation (rTMS). Only a handful of studies have attempted to promote cognitive functioning after stroke with rTMS. These studies exclusively used a one-size-fits-all approach, which had limited success, as post-stroke cognitive deficits are highly variable. We propose a two-step personalized treatment strategy to identify targets for therapeutic TMS for cognitive rehabilitation after stroke. Step one consits of identification of personalized TMS targets by measuring fMRI activity during a representative cognitive task. In step two, TMS disruption is used to temporarily disrupt activity in the targeted brain region to investigate causal involvement of a brain area in cognitive task performance.

Objective: To validate a proof-of-concept to identify personalized targets for therapeutic TMS for cognitive rehabilitation after stroke.

Study design: A prospective mechanistic intervention study.

Study population: 10 healthy individuals and 15 stroke patients with cognitive impairment

Intervention: Active and sham TMS disruption of personalized targets

Main study endpoints: The n-back test

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. First-ever ischemic stroke or intracerebral haemorrhage in a cerebral hemisphere or the brainstem;
3. Cognitive impairment based on assessment by the treating rehabilitation physician.
4. Able to perform n-back task at inclusion.
5. Inclusion possible within 10 weeks after stroke onset;
6. Signed informed consent.

Exclusion Criteria:

1. Known cognitive impairment prior to stroke onset;
2. Absolute contra-indication to TMS: Magnetic sensitive objects implanted in the head or neck area (e.g. cochlear implants, implanted neurostimulator, pacemaker or defibrillator, metal splinters, metal fragments or metal clips), history of epilepsy, pregnancy or other contra-indications that may potentially be harmful as determined by the treating rehabilitation physician;
3. Incompetence or severe impairments that can impede study participation as determined by the treating rehabilitation physician (i.e. extreme fatigue, severe communication deficits);
4. Life expectancy shorter than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in n-back test performance | during TMS disruption

IPD SHARING:
Plan to Share IPD: No
Anonymized patient data can be made available on request